CLINICAL TRIAL: NCT00842387
Title: Evaluation Study of a Management Strategy for Gastroesophageal Reflux Disease (GERD)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Rick Lones, European Medical Affairs Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-GEU-DUM-2008/1
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Reflux; Heartburn; Regurgitation; Esophagitis
Keywords: gastroesophageal reflux disease; reflux, heartburn; regurgitation; acid control; PPI; antiacid; primary care; esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with symptoms suggestive of GERD, managed according to a new structured and implemented pathway
- 2: Patients with symptoms suggestive of GERD, managed according to usual clinical practice.

SUMMARY:
The aim of this project is to compare the GERD clinical outcomes in patients where a structured pathway using the GerdQ questionnaire is implemented compared with the clinical outcomes of those treated without this implementation.

This is a European project with 5 participating countries (Austria, Italy, Norway, Spain and Sweden). Due to different characteristics regarding the actual management of this disease in the 5 countries, each country had the flexibility to introduce design differences and changes in the study protocol.

DETAILED DESCRIPTION:
In Norway, it is developed as a clinical trial where a new structured pathway in the diagnosis and treatment of GERD is compared to the ordinary clinical pathway consisting of the endoscopic/pH-metry approach in patients referred from primary care to GI specialists.

In Italy, it is a PCP-level, cluster randomized, controlled trial comparing a structured clinical pathway versus usual care in patients with GERD. The implementation consists of training sessions on the clinical pathway with the selected PCPs (Implementation Group).

In Sweden, it is a cluster-randomised interventional study performed within daily clinical practice for the purpose of assessing the effect of the implementation of the structured clinical pathway in patients identified as having GERD. The participating PCCs will be randomised (1:1) to implement the structured clinical pathway or handling the patients according to local clinical routines.

In Austria and Spain, it is a cluster-randomized study to be developed within daily clinical practice for the purpose of assessing the effect of the implementation of the structured clinical pathway on GERD patients . The evaluation study will take place subsequent to a prior implementation of a clinical pathway. The implementation consists of a detailed explanation by training-materials about the clinical pathway in a selected randomized pool of PCCs. The implementation that will be evaluated is outside of the study procedures; it is the physician's decision whether to apply it or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with symptoms suggestive of GERD (heartburn or regurgitation as prevailing symptoms) of any severity
* Patient able to understand and complete the questionnaires

Exclusion Criteria:

* Alarm symptoms (Dysphagia/odynophagia, anorexia, anaemia, unintentional weight loss, abdominal mass, upper GI bleeding)
* If the patient is participating in any clinical trial, he/she cannot take part on this study
* Any condition that, in the investigator's opinion, makes the patient's participation in the study difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptoms suggestive of GERD.
Sampling Method: Probability Sample
Enrollment: 2370 (Estimated)
Dates: Start 2009-01; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Control of symptoms based on results of GerdQ, need of treatment change and % of patients requiring referral to a specialist (Austria and Italy). | up to 8 weeks
Treatment response and symptomatic control (Norway) | up to 8 weeks
Symptom relief and patient satisfaction with treatment (Spain) | up to 8 weeks
Symptom relief measured by RDQ (Sweden) | 5 months +/- 4 weeks

SECONDARY OUTCOMES:
Use and consumption of healthcare resources (all countries). Physicians adherence to the clinical pathway (Austria, Spain) and intrinsic characteristics of the physicians/PCC that may affect this adherence (Austria) | Up to 8 weeks, except for Sweden: 5 months +/- 4 weeks
Percentage of patients referred to specialists (Spain). Health status based on EQ-5D measure (Norway, Sweden). Work productivity based on the WPAI-GERD questionnaire (Norway, Sweden) | Up to 8 weeks, except for Sweden: 5 months +/- 4 weeks
Sweden: Persisting symptoms according to GerdQ, Treatment changes, Reason(s) for the patient consultation at visit 1. To explore other GERD related symptoms, To describe patients' experience of treatment/care given during the study. | 5 months +/- 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mónica Tafalla, MD, Study Director — Medical DepartmentAstraZeneca Spain
Locations (66):
- Austria (30):
  - Research Site, Amstetten
  - Research Site, Baden
  - Research Site, Bludenz
  - Research Site, Bregenz
  - Research Site, Feldbach
  - Research Site, Gmunden
  - Research Site, Graz
  - Research Site, Groß-Gerungs
  - Research Site, Innsbruck
  - Research Site, Kitzbühel
  - Research Site, Klagenfurt
  - Research Site, Krems
  - Research Site, Kufstein
  - Research Site, Leibnitz, Styria
  - Research Site, Leoben
  - Research Site, Linz
  - Research Site, Mattersburg
  - Research Site, Mistelbach
  - Research Site, Mürzzuschlag
  - Research Site, Neunkirchen
  - Research Site, Neusiedl
  - Research Site, Perg
  - Research Site, Sankt Veit im Pongau
  - Research Site, Schwaz
  - Research Site, Steyr
  - Research Site, Villach
  - Research Site, Vöcklabruck
  - Research Site, Völkermarkt
  - Research Site, Wels
  - Research Site, Zell
- Research Site, Brescia, Italy
- Norway (12):
  - Research Site, Arendal
  - Research Site, Ålesund
  - Research Site, Bergen
  - Research Site, Bodø
  - Research Site, Haugesund
  - Research Site, Kristiansund
  - Research Site, Levanger
  - Research Site, Molde
  - Research Site, Mosjøen
  - Research Site, Orkdal
  - Research Site, Oslo
  - Research Site, Tynset
- Research Site, Valencia, Spain
- Sweden (22):
  - Research Site, Arlöv
  - Research Site, Dalby
  - Research Site, Falköping
  - Research Site, Farsta
  - Research Site, Gothenburg
  - Research Site, Helsingborg
  - Research Site, Karlshamn
  - Research Site, Kristianstad
  - Research Site, Kungsängen
  - Research Site, Luleå
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Munkedal
  - Research Site, Nordstan(Goteborg)
  - Research Site, Partille
  - Research Site, Piteå
  - Research Site, Skanör
  - Research Site, Solna
  - Research Site, Södertälje
  - Research Site, Stockholm
  - Research Site, Trollhättan
  - Research Site, Vännäs

REFERENCES:
- [Derived] Bergquist H, Agreus L, Tillander L, Johnsson F, Sorngard H, Sjostedt S, Hellstrom PM. Structured diagnostic and treatment approach versus the usual primary care approach in patients with gastroesophageal reflux disease: a cluster-randomized multicenter study. J Clin Gastroenterol. 2013 Aug;47(7):e65-73. doi: 10.1097/MCG.0b013e31827d7782. PMID 23426452
- [Derived] Jonasson C, Moum B, Bang C, Andersen KR, Hatlebakk JG. Randomised clinical trial: a comparison between a GerdQ-based algorithm and an endoscopy-based approach for the diagnosis and initial treatment of GERD. Aliment Pharmacol Ther. 2012 Jun;35(11):1290-300. doi: 10.1111/j.1365-2036.2012.05092.x. Epub 2012 Apr 18. PMID 22510027